CLINICAL TRIAL: NCT07306221
Title: Effect of Visual-Guided Balance Training on Knee Motor Function and Biomechanical Characteristics After ACL Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M20250822
Record Dates: First submitted 2025-11-20; First posted 2025-12-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament injuries; Visual-guided balance training; gait; ACLR; reconstruction of anterior cruciate ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy control group (No Intervention): The main focus is on conducting a comparative analysis of health conditions based on the analysis of motor functions.
- Traditional group (Active Comparator): Based on the conventional standardized rehabilitation procedures, additional general balance training content is added.
  Interventions: Other: Traditional group
- Intervention group (Experimental): Based on the conventional standardized rehabilitation program, add the content of visual-guided balance training
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Traditional group — Based on the traditional standardized rehabilitation program, additional universal balance training content has been added. Starting from the 5th week after the surgery and continuing until the 14th week, three times a week for a total of 10 weeks, the training duration was one and a half hours each time.
  Arms: Traditional group
Other: Intervention Group — Based on the conventional standardized rehabilitation program, add the content of visual-guided balance training.Starting from the 5th week after the surgery and continuing until the 14th week, three times a week for a total of 10 weeks, the training duration was one and a half hours each time.
  Arms: Intervention group

SUMMARY:
This study aims to investigate the improvement effect of visual-guided balance training on the knee joint function and gait performance of patients after ACLR, and to clarify the advantages of this training program compared to conventional rehabilitation training; at the same time, by including healthy individuals as the control group, it quantifies the differences in knee joint function and gait performance between patients after ACLR and healthy individuals, to verify whether visual-guided balance training can more effectively narrow the functional gap between patients after ACLR and healthy individuals, and promote the recovery of patients' knee joint function and gait closer to the healthy level. Ultimately, it provides scientific theoretical basis and practical guidance for the optimization of the rehabilitation plan after ACLR, and helps patients achieve comprehensive and high-quality recovery.

DETAILED DESCRIPTION:
In this randomized controlled clinical study, patients with primary unilateral anterior cruciate ligament rupture were included. Starting from the 5th week after surgery, in addition to the standardized rehabilitation training content, the traditional group added general balance training, and the intervention group added visual guidance balance training. The analysis was conducted through movement function tests and evaluations, with the healthy group included as the control. The impact of visual guidance balance training on the movement function and biomechanical characteristics after ACLR was explored.

ELIGIBILITY:
Inclusion criteria for patients:

1. Age between 18 and 45 years old;
2. Body Mass Index (BMI) ranging from 18.5 kg/m² to less than 35 kg/m²;
3. First unilateral ACL rupture and reconstruction surgery performed at this hospital;
4. Autologous hamstring tendon transplantation;
5. No or only minor injury to the meniscus, posterior cruciate ligament, medial collateral ligament or lateral collateral ligament;
6. Voluntary participation in this study and signing of informed consent form.

Exclusion criteria for patients:

1. Patients who underwent ACL reconstruction more than one year after the injury;
2. Patients with severe injuries to the posterior cruciate ligament, medial collateral ligament or lateral collateral ligament (more than grade I; grade II is partial tear, thickening and tortuosity of the ligament, partial fiber interruption, and swelling of the surrounding soft tissues; grade III is complete rupture). ； Combined with severe meniscus tear;
3. Has a history of previous knee surgery, such as meniscus repair, ligament reconstruction, joint replacement, joint cleaning, etc.;
4. Has other knee joint diseases, such as: knee osteoarthritis, knee joint tumor, rheumatoid arthritis, tuberculosis, knee joint infection or inflammatory diseases, fracture, dislocation or other bone injuries, etc.;
5. Severe heart, lung, brain diseases or liver and kidney dysfunction, and visual and cognitive impairments.

Inclusion criteria for the healthy control group

1. Age 18-45 years old;
2. Body Mass Index (BMI) ≥ 18.5 kg/m2 and < 35 kg/m2;
3. No surgical history, injury history, or chronic joint diseases of the lower extremities;
4. No visual, cognitive impairments or neurological diseases;
5. No trauma or diseases that cause abnormal gait. Exclusion criteria

1. Poor compliance of the subject; 2. The subject withdraws the informed consent form; 3.The subject requests to terminate the study or is unable to complete all the trials for some reason; 4. The investigator believes that the subject's continued participation in the trial may cause significant adverse effects on their physical condition; 5. The ethics review committee decides to terminate the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Vicon 3D Gait Testing | Preoperative baseline; 14 weeks after the operation; 6 months after the operation
  The subjects first underwent a static test, and then chose to perform tests of slow jogging, walking and single-leg balance at their own pace. Observe the three-dimensional plane joint angles（degree) of each joint in the lower limbs.
Vicon 3D Gait Testing | Preoperative baseline; 14 weeks after the operation; 6 months after the operation
  The subjects first underwent a static test, and then chose to perform tests of slow jogging, walking and single-leg balance at their own pace. Observe the three-dimensional plane joint torques (BW×BH）of each joint in the lower limbs.
Vicon 3D Gait Testing | Preoperative baseline; 14 weeks after the operation; 6 months after the operation
  After a static trial, participants performed self-paced tests of slow jogging, walking, and single-leg balance while three-dimensional ground reaction forces （BW)at each lower-limb joint were recorded.
isokinetic muscle strength | Preoperative baseline;14 weeks after the operation; 6 months after the operation
  This isokinetic muscle strength test selected two angular velocities: 60°/second (slow speed) and 180°/second (medium speed). Observe the relative peak torque （ N·m/kg）of the quadriceps and hamstring muscles.
isokinetic muscle strength | Preoperative baseline;14 weeks after the operation; 6 months after the operation
  This isokinetic muscle strength test selected two angular velocities: 60°/second (slow speed) and 180°/second (medium speed).Observe the limb symmetry index（%） of the quadriceps and hamstring muscles.
isokinetic muscle strength | Preoperative baseline;14 weeks after the operation; 6 months after the operation
  This isokinetic muscle strength test selected two angular velocities: 60°/second (slow speed) and 180°/second (medium speed).Observe the hamstring-to-quadriceps peak-torque ratio (H/Q).
Imoove Balance Training Tester | Preoperative baseline; 4 weeks after the operation; 14 weeks after the operation; 6 months after the operation
  The dynamic balance ability of the subjects was evaluated. The main observations included the imbalance percentage, the score of the green target, coordination, stability, distribution balance, and the total score. The score ranged from 0 to 100, with a higher score being better.

SECONDARY OUTCOMES:
Lysholm Knee Joint Scoring Scale | Preoperative baseline; 4 weeks after the operation; 14 weeks after the operation; 6 months after the operation
  The Lysholm Knee Joint Scoring Scale is a tool used to evaluate the function of the knee joint and to monitor the rehabilitation process after knee joint injury or surgery. The score ranges from 0 to 100, with a higher score indicating better recovery of knee joint function. The score ranges from 0 to 100.
International Knee Documentation Committee Knee Assessment Scale | Preoperative baseline; 4 weeks after the operation; 14 weeks after the operation; 6 months after the operation
  The International Knee Documentation Committee Knee Assessment Scale is a comprehensive tool used to evaluate knee joint function. It aims to provide standardized assessment for patients with knee joint injuries or after surgery, with a score range of 0 to 100. The higher the score, the better.
Visual Analogue Score | Preoperative baseline; 4 weeks after the operation; 14 weeks after the operation; 6 months after the operation
  It is mainly used to rate the degree of patient's pain, with scores ranging from 0 to 10. The lower the score, the better.
Tampa Scale for Kinesiophobia-11 | Preoperative baseline; 4 weeks after the operation; 14 weeks after the operation; 6 months after the operation
  TSK-11 (Tampa Scale for Kinesiophobia-11, a simplified version of the Tampa Scale for Kinesiophobia) is a tool used to assess an individual's fear of movement/body activity (kinesiophobia). It consists of 11 items, with a total score ranging from 11 to 44; the scoring rule is as follows: ≤ 26 points indicate no significant kinesiophobia, while > 26 points indicate the presence of kinesiophobia, and the higher the score, the greater the fear of movement and the more severe the avoidance tendency.
ACL Return to Sport after Injury scale | Preoperative baseline; 4 weeks after the operation; 14 weeks after the operation; 6 months after the operation
  The ACL Recovery Sport Readiness Index (ACL-RSI) is a scale used to assess the psychological readiness of patients with anterior cruciate ligament (ACL) injury/reconstruction to return to sports. This scale consists of 12 items and is scored on a scale of 0 to 100. The higher the score, the better.

CONTACTS AND LOCATIONS:
Overall Officials: ren shuang, doctor, Study Chair — Be affiliated with the organization
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No